CLINICAL TRIAL: NCT07407543
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Doses, Dose-escalation Phase 1 Clinical Trial to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SRN001 in Healthy Korean and Caucasian Adult Males
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SRN001 in Healthy Korean and Caucasian Adult Males
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: siRNAgen Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRN001-CA-25001A
Record Dates: First submitted 2026-01-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cohort1 Drug: SRN001 45mg (Experimental): cohort1 Drug: SRN001 45mg
  Interventions: Drug: SRN001
- cohort2 Drug: SRN001 90mg (Experimental): cohort2 Drug: SRN001 90mg
  Interventions: Drug: SRN001
- cohort3 Drug: SRN001 180mg (Experimental): cohort3 Drug: SRN001 180mg
  Interventions: Drug: SRN001
- Placebo Comparator (Placebo Comparator): Participants receive placebo (0.9% sodium chloride, normal saline)
  Interventions: Drug: 0.9% sodium chloride (normal saline)

INTERVENTIONS:
Drug: SRN001 — SRN001 is an investigational drug administered at doses of 45 mg, 90 mg, or 180 mg depending on cohort.
  Arms: cohort1 Drug: SRN001 45mg; cohort2 Drug: SRN001 90mg; cohort3 Drug: SRN001 180mg
Drug: 0.9% sodium chloride (normal saline) — 0.9% sodium chloride solution administered as placebo control.
  Arms: Placebo Comparator

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of repeated doses of SRN001 in healthy adult volunteers.

DETAILED DESCRIPTION:
SRN001 is a novel small interfering RNA (siRNA) drug being developed to treat fibrosis using Self Assembled Micelle inhibitory ribonucleic acid (SAMiRNA™) technology. Amphiregulin (AREG) is a growth factor involved in fibroblast proliferation and myofibroblast transformation which is the hallmark of fibrosis in lung and kidney tissues. AREG is a downstream gene overexpressed by Transforming growth factor-β (TGF-β) during fibrosis, promoting fibroblast to myofibroblast transition (FMT). SRN001 is designed to downregulate generating amphiregulin by RNA interference (RNAi). The goal of this clinical trial is to evaluate safety, tolerability, pharmacokinetics and pharmacodynamics of SRN001 in healthy Korean and Caucasian adult males.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Korean or Caucasian male volunteers aged 19 to 60 years at the time of screening.
2. Those who weighed 50.0 kg or more at the time of screening and had a body mass index (BMI) between 18.5 kg/m2 and 29.9 kg/m2.

   Body mass index (BMI, kg/m2) = weight (kg) / {height (m2)} 2
3. Those whose screening results showed a serum amphiregulin concentration of 100 pg/mL or higher.
4. Those who voluntarily agreed to participate in this clinical trial after receiving a thorough explanation and fully understanding the clinical trial. Those who decided to participate and gave written consent to comply with the precautions.

Exclusion Criteria:

1. Those with or have a history of clinically significant diseases of the hepatobiliary system (severe liver failure, viral hepatitis, etc.), kidney (severe renal failure, etc.), nervous system, immune system, respiratory system, digestive system, endocrine system, hematological/oncological system, cardiovascular system (heart failure, torsades de pointes, etc.), urinary system, psychiatric system (mood disorder, obsessive-compulsive disorder, etc.), or sexual dysfunction.
2. Those with a history of hypersensitivity to RNA drugs or other drugs (aspirin, antibiotics, etc.) or a history of clinically significant hypersensitivity reactions (atopy, asthma, etc.).
3. Those with a positive serum test result (hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test, syphilis test).
4. Those with a history of drug abuse or a positive urine drug screening test for drugs of abuse.
5. Those who were screened in a sitting position after resting for at least 3 minutes. Those who exhibited the following values in measured vital signs:

   * Systolic blood pressure < 80 mmHg or ≥ 140 mmHg
   * Diastolic blood pressure < 45 mmHg or ≥ 90 mmHg
   * Pulse < 45 bpm or > 100 bpm
   * Body temperature < 35.5 ℃ or > 37.7 ℃
6. Those who exhibited the following values or clinically significant abnormal rhythm findings on the electrocardiogram (12-lead ECG) during the screening test:

   -QTcF > 450 msec
7. Those who exhibited one or more of the following results in clinical laboratory tests during the screening test, including additional tests:

   * AST (SGOT) or ALT (SGPT) > 60 IU/L
   * Estimated glomerular filtration rate (CKD-EPI equation) < 60 mL/min/1.73 m2
8. Those who have taken any prescription drugs or herbal medicines within two weeks prior to the scheduled first administration of the investigational drug, or have taken any over-the-counter drugs, health functional foods including liver function supplements, or vitamin preparations within one week (however, at the investigator's discretion, subjects may be selected as subjects if other conditions are appropriate) or are expected to take such drugs.
9. Those who have taken drug-metabolizing enzyme inducers such as barbiturates or drug metabolism inhibitors such as clarithromycin within one month prior to the scheduled first administration of the investigational drug.
10. Those who have participated in another clinical trial (including bioequivalence trials) and received the investigational drug within six months prior to the scheduled first administration of the investigational drug.
11. Those who have donated whole blood within two months prior to the scheduled first administration of the investigational drug, or have donated blood components within one month prior to the scheduled first administration of the investigational drug, or have received a blood transfusion.
12. Smokers (however, subjects may be selected as subjects if they quit smoking three months prior to the scheduled first administration of the investigational drug) or those who are unable to quit smoking until the completion of the clinical trial.
13. Those who have continuously consumed alcohol (21 units/week, 1 unit = 10 g of pure alcohol) or cannot abstain from alcohol from 3 days before the scheduled first dose of the investigational drug until the end of the clinical trial.
14. Those who have continuously consumed excessive caffeine (more than 5 units/day, 1 unit = 80 mg of caffeine) or cannot abstain from consuming caffeinated foods and beverages (coffee, tea (black tea, green tea, etc.), carbonated beverages, coffee drinks, coffee milk, tonic drinks, energy drinks, etc.) from 3 days before the scheduled first dose of the investigational drug until the end of the clinical trial.
15. Those who cannot abstain from consuming grapefruit (grapefruit), grapefruit juice, or grapefruit-containing foods from 3 days before the scheduled first dose of the investigational drug until the end of the clinical trial.
16. Those who have unusual eating habits (e.g., consuming more than 1 L of grapefruit juice per day) or cannot consume the standardized diet provided by the clinical trial center during their hospitalization.
17. Those who use their own condoms from 3 days before the scheduled first dose of the investigational drug until the end of the clinical trial. Women of childbearing potential (spouse or partner) who do not consent to a contraceptive method considered highly effective.

    [Contraceptive methods considered highly effective]
18. Those who do not agree to refrain from donating sperm from 3 days prior to the scheduled first dose of the investigational drug until the end of the clinical trial.
19. Those whom the investigator determines to be unsuitable for clinical trial participation for reasons other than those listed above.

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From first dose through end of study (up to 114 days)
  Number of participants experiencing one or more TEAEs during the study period.
Number of participants with serious adverse events (SAEs) | From first dose through end of study (up to 114 days)
  Number of participants with SAEs as defined in protocol.
Number of participants with clinically significant abnormal laboratory results | From first dose through end of study (up to 114 days)
  Counts of clinically significant abnormal lab tests during study.
Maximum Observed Plasma Concentration (Cmax) of SRN001 | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose)
  Maximum observed plasma concentration (Cmax) following IV administration of SRN001.
Time to Maximum Plasma Concentration (Tmax) of SRN001 | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose) Post-dose samples (Day 1 and Day 29): 0 (end of infusion), 10, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 6, 12, 24, and 48 hours after dosing
  Time to reach maximum observed plasma concentration following IV administration.
Area Under the Curve from time zero to last measurable concentration (AUClast) | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose) Post-dose samples (Day 1 and Day 29): 0 (end of infusion), 10, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 6, 12, 24, and 48 hours after dosing
  AUClast of SRN001 plasma concentration versus time curve.
Area Under the Plasma Concentration-Time Curve over the Dosing Interval (AUCtau) of SRN001 | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose) Post-dose samples (Day 1 and Day 29): 0 (end of infusion), 10, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 6, 12, 24, and 48 hours after dosing
  AUCtau will be calculated as the area under the plasma concentration versus time curve over one complete dosing interval following multiple escalating intravenous doses of SRN001.
Terminal Half-Life (t½) of SRN001 | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose) Post-dose samples (Day 1 and Day 29): 0 (end of infusion), 10, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 6, 12, 24, and 48 hours after dosing
  Terminal elimination half-life (t½) will be calculated from the plasma concentration-time profile at steady state following multiple doses.
Clearance (CL) of SRN001 | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose) Post-dose samples (Day 1 and Day 29): 0 (end of infusion), 10, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 6, 12, 24, and 48 hours after dosing
  Systemic clearance (CL) will be determined from non-compartmental analysis of plasma concentrations at steady state after multiple dosing.
Apparent Volume of Distribution (Vz) of SRN001 | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose) Post-dose samples (Day 1 and Day 29): 0 (end of infusion), 10, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 6, 12, 24, and 48 hours after dosing
  Apparent volume of distribution (Vz) will be calculated from plasma concentration data at steady state following multiple doses.
Time to Maximum Observed Plasma Concentration at Steady State (Tmax,ss) of SRN001 | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose) Post-dose samples (Day 1 and Day 29): 0 (end of infusion), 10, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 6, 12, 24, and 48 hours after dosing
  Time to reach maximum observed plasma concentration at steady state following multiple intravenous doses.
Maximum Observed Plasma Concentration at Steady State (Cmax,ss) of SRN001 | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose) Post-dose samples (Day 1 and Day 29): 0 (end of infusion), 10, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 6, 12, 24, and 48 hours after dosing
  Maximum observed plasma concentration at steady state following multiple intravenous doses.
Minimum Observed Plasma Concentration at Steady State (Cmin,ss) of SRN001 | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose) Post-dose samples (Day 1 and Day 29): 0 (end of infusion), 10, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 6, 12, 24, and 48 hours after dosing
  Minimum observed plasma concentration at steady state following multiple doses.
Average Plasma Concentration at Steady State (Cavg,ss) of SRN001 | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose) Post-dose samples (Day 1 and Day 29): 0 (end of infusion), 10, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 6, 12, 24, and 48 hours after dosing
  Average plasma concentration at steady state following multiple intravenous doses.
Trough Plasma Concentration at Steady State (Ctrough) of SRN001 | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose) Post-dose samples (Day 1 and Day 29): 0 (end of infusion), 10, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 6, 12, 24, and 48 hours after dosing
  Plasma concentration just prior to the next dose at steady state following multiple dosing.
Area Under the Plasma Concentration-Time Curve over the Dosing Interval at Steady State (AUCtau,ss) of SRN001 | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose) Post-dose samples (Day 1 and Day 29): 0 (end of infusion), 10, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 6, 12, 24, and 48 hours after dosing
  AUCtau,ss will be calculated over one dosing interval at steady state following multiple intravenous doses.
Peak-to-Trough Fluctuation (PTF) of SRN001 at Steady State Description: Peak-to-trough fluctuation in plasma concentration at steady state, defined as (Cmax,ss - Cmin,ss)/Cavg,ss. | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose) Post-dose samples (Day 1 and Day 29): 0 (end of infusion), 10, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 6, 12, 24, and 48 hours after dosing
  Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose)
Accumulation Ratio (R) of SRN001 at Steady State | Pre-dose samples: Day 1, Day 15, and Day 29 (pre-dose) Post-dose samples (Day 1 and Day 29): 0 (end of infusion), 10, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 6, 12, 24, and 48 hours after dosing
  Accumulation ratio (R) comparing exposure at steady state with that after the first dose (e.g., based on Cmax or AUC).

OTHER OUTCOMES:
Changes in Serum Amphiregulin Concentration | Changes from baseline in circulating amphiregulin concentrations will be evaluated using 11 blood sampling time points, including pre-dose, early post-dose, and follow-up assessments.
  Baseline to post-study visit (pre-dose on Days 1, 15, and 29; post-dose on Days 1 and 29 at 2 and 12 hours; and at Days 43, 57, 85, and end-of-study)
Changes in PBMC LPS-Stimulated Amphiregulin Levels | Baseline to Day 29 (pre-dose on Days 1, 15, and 29; post-dose at 2 and 24 hours on Days 1 and 29)
  PBMCs collected will be stimulated ex vivo with LPS, and increases in amphiregulin concentrations relative to baseline will be measured across 7 sampling time points.
Changes in Urine Albumin-to-Creatinine Ratio (uACR) | Day 1 to 48 hours post-dose on Day 29 (pre-dose and 0-3, 3-6, 6-12, 12-24, and 24-48 hours post-dose)
  Changes from baseline in urine ACR (albumin/creatinine ratio) will be assessed.
Changes in Serum Inflammatory Cytokines (IFN-γ, IL-6, IL-1β, TNFα) | Baseline to Day 29 (pre-dose on Days 1, 15, and 29; post-dose 1, 6, and 12 hours on Days 1, 15, and 29)
  Changes from baseline in serum concentrations of IFN-γ, IL-6, IL-1β, and TNFα will be assessed at 12 time points, including pre-dose and multiple post-dose intervals.
Incidence of Anti-SRN001 Antibody Formation | Baseline to end-of-study visit (pre-dose on Days 1, 15, and 29; and follow-up on Day 57 and post-study visit)
  Presence of anti-SRN001 antibodies will be evaluated. If antibody positivity is detected, antibody titers will be quantified across five serum sampling time points.
Maximum Observed SRN001 Concentration in PBMCs (Cmax) | 30 Minutes Post-Dose on Day 1
  Cmax is the maximum observed SRN001 concentration in peripheral blood mononuclear cells following drug administration.
Area Under PBMC Concentration-Time Curve (AUCtau) | Sampling up to 12 Hours Post-Dose on Day 1
  AUCtau is the area under the plasma concentration versus time curve over the dosing interval for SRN001 in PBMCs.
Area Under PBMC Concentration-Time Curve from Time Zero to Last Measurement (AUClast) | Sampling up to 12 Hours Post-Dose on Day 1
  AUClast is the area under the PBMC concentration versus time curve from predose until the last quantifiable concentration.
Maximum Observed SRN001 Concentration in PBMCs at Steady State (Cmax,ss) | 30 Minutes Post-Dose on Day 29
  Cmax,ss is the maximum SRN001 concentration observed in PBMCs at steady state after multiple doses.
Area Under PBMC Concentration-Time Curve at Steady State (AUCtau,ss) | Sampling up to 12 Hours Post-Dose on Day 29
  AUCtau,ss is the area under the PBMC concentration versus time curve over one dosing interval at steady state.
Accumulation Ratio of SRN001 in PBMCs (R) | From Predose on Day 1 and Predose on Day 29
  Accumulation ratio is the ratio of exposure at steady state (AUCtau,ss) relative to single dose exposure (AUCtau).
PBMC-to-Plasma Concentration Ratio of SRN001 at Steady State | Sampling at 30 Minutes Post-Dose on Day 29
  Ratio of SRN001 concentration in PBMCs versus plasma at steady state.
Change in Serum Amphiregulin Concentration from Baseline to 2 Hours Post-Dose on Day 1 | Baseline and 2 Hours Post-Dose on Day 1
  Change from baseline in circulating amphiregulin concentration through 2 hours after dosing on Day 1, as measured in blood samples.
Change in Serum Amphiregulin Concentration from Baseline to 12 Hours Post-Dose on Day 1 | Baseline and 12 Hours Post-Dose on Day 1
  Change from baseline in circulating amphiregulin concentration through 12 hours after dosing on Day 1.
Change in Serum Amphiregulin Concentration from Baseline to Predose on Day 15 | Baseline and Predose on Day 15
  Change from baseline in circulating amphiregulin concentration measured prior to dosing on Day 15.
Change in Serum Amphiregulin Concentration from Baseline to Predose on Day 29 | Baseline and Predose on Day 29.
  Change from baseline in circulating amphiregulin concentration measured prior to dosing on Day 29.
Change in Serum Amphiregulin Concentration from Baseline to Predose on Day 43 | Baseline and Predose on Day 43
  Change from baseline in circulating amphiregulin concentration measured at predose (0 hour) on Day 43.
Change in Serum Amphiregulin Concentration from Baseline to Predose on Day 57 | Baseline and Predose on Day 57
  Change from baseline in circulating amphiregulin concentration measured at predose (0 hour) on Day 57.
Change in Serum Amphiregulin Concentration from Baseline to Predose on Day 85 | Baseline and Predose on Day 85
  Change from baseline in circulating amphiregulin concentration measured at predose (0 hour) on Day 85.
Change in Serum Amphiregulin Concentration from Baseline to End-of-Study Visit (Post-Study Visit) | Baseline and Day 111-114
  Change from baseline in circulating amphiregulin concentration measured at the post-study visit conducted between Day 111 and Day 114.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Yoon PO, Park JW, Lee CM, Kim SH, Kim HN, Ko Y, Bae SJ, Yun S, Park JH, Kwon T, Kim WS, Lee J, Lu Q, Kang HR, Cho WK, Elias JA, Yang JS, Park HO, Lee K, Lee CG. Self-assembled Micelle Interfering RNA for Effective and Safe Targeting of Dysregulated Genes in Pulmonary Fibrosis. J Biol Chem. 2016 Mar 18;291(12):6433-46. doi: 10.1074/jbc.M115.693671. Epub 2016 Jan 27. PMID 26817844
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26817844/